CLINICAL TRIAL: NCT06600464
Title: Is There a Relationship Between Ultrasound Findings of Thumb Muscles and Grip Strength in Addition to Pain Threshold in Thumb Carpometacarpal Osteoarthritis
Brief Title: Ultrasound Findings of Thumb Muscles in 1st Carpometacarpal Osteoarthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gulcanozturk1984
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthrosis; Ultrasound
Keywords: osteoarthrosis; ultrasound; thenar muscles
MeSH Terms: conditions — Osteoarthritis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with various stages of 1st carpometacarpal (CMC) joint osteoarthritis (OA) were assessed using standard radiographs based on the Modified Eaton Litter classification
  Interventions: Diagnostic Test: Ultrasound; Other: Assessment of Muscle Strength in Both Hands; Other: Assessment of Pain Threshold
- Group 2: In the healthy control group, subjects were matched based on age and hand dominance
  Interventions: Diagnostic Test: Ultrasound; Other: Assessment of Muscle Strength in Both Hands; Other: Assessment of Pain Threshold

INTERVENTIONS:
Diagnostic Test: Ultrasound — The thickness of the thenar eminence muscles (longitudinal thickness of the first dorsal interosseous muscle (FDI), abductor pollicis brevis (APB), and opponens pollicis (OPP)) was measured using musculoskeletal ultrasound.
Other: Assessment of Muscle Strength in Both Hands — Muscle strength in both hands was evaluated using grip strength measured with a dynamometer (Jamar Hydraulic Hand Dynamometer, Nottinghamshire, UK)
Other: Assessment of Pain Threshold — Pressure pain threshold (PPT) for painful and non-painful finger joints was assessed using a hand-held algometer

SUMMARY:
Carpometacarpal (CMC) joint osteoarthritis is a disorder that is estimated to affect more than one-third of postmenopausal women, leading to decreased muscle strength, reduced joint range of motion, and pain.The pathogenesis of thumb CMC osteoarthritis involves complex interactions between biomechanical forces, genetic predisposition, hormonal changes, repetitive microtrauma, and aging. An important factor in the progression of carpometacarpal osteoarthritis is the loss of joint stability provided by the surrounding muscles (2). The common methods for diagnosing thumb CMC OA is plain radiographs and clinical examinations. However, radiographs are unable to assess the role of surrounding structures, including muscles and ligaments.

Ultrasound is a cost-effective, radiation-free, and easily applicable imaging method.

DETAILED DESCRIPTION:
In this cross-sectional study, patients with various stages of 1st carpometacarpal (CMC) joint osteoarthritis (OA) were assessed using standard radiographs based on the Modified Eaton Litter classification. Postmenopausal women with clinical and/or radiological evidence of 1st CMC OA will be included (Group 1). In the healthy control group, subjects will be matched based on age and hand dominance (Group 2). Demographic information including age, sex, height, weight, body mass index (BMI, kg/m²), dominant hand, and symptom duration (in months) will recorded. Pain levels will be assessed using the Visual Analogue Scale (VAS).The thickness of the thenar eminence muscles (longitudinal thickness of the first dorsal interosseous muscle (FDI), abductor pollicis brevis (APB), and opponens pollicis (OPP)) was measured using musculoskeletal ultrasound. Muscle strength in both hands will be evaluated using grip strength measured with a dynamometer . Pressure pain threshold (PPT) for painful and non-painful finger joints will be assessed using a hand-held algometer

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women with clinical and/or radiological evidence of 1st CMC OA

Exclusion Criteria:

* De Quervain's tenosynovitis, flexor carpi radialis tendon pathology, and carpal tunnel syndrome, as well as those with hand trauma or hand surgery within the past year, had received steroid and local anesthetic injections into the 1st CMC joint within the last 3 months, or had connective tissue disorders, rheumatologic, or autoimmune diseases

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with clinical and/or radiological evidence of 1st CMC OA
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrasound | 1 day
  The thickness of the thenar eminence muscles (longitudinal thickness of the first dorsal interosseous muscle (FDI), abductor pollicis brevis (APB), and opponens pollicis (OPP)) was measured using musculoskeletal ultrasound.
Assessment of Muscle Strength in Both Hands | 1 day
  Participants were seated in a standardized position with their elbows flexed at 90°. Muscle strength in both hands was evaluated using grip strength measured with a dynamometer (Jamar Hydraulic Hand Dynamometer, Nottinghamshire, UK)
Assessment of Pain Threshold | 1 day
  Pressure pain threshold (PPT) for painful and non-painful finger joints was assessed using a hand-held algometer (FPIX25, with a 1 cm² flat rubber probe).

CONTACTS AND LOCATIONS:
Locations (1):
- Gulcan Ozturk, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mohseny B, Nijhuis TH, Hundepool CA, Janssen WG, Selles RW, Coert JH. Ultrasonographic quantification of intrinsic hand muscle cross-sectional area; reliability and validity for predicting muscle strength. Arch Phys Med Rehabil. 2015 May;96(5):845-53. doi: 10.1016/j.apmr.2014.11.014. Epub 2014 Dec 4. PMID 25482051
- [Result] Pickrell BB, Eberlin KR. Thumb Basal Joint Arthritis. Clin Plast Surg. 2019 Jul;46(3):407-413. doi: 10.1016/j.cps.2019.02.010. PMID 31103085
- See also: Pickrell BB, Eberlin KR. Thumb Basal Joint Arthritis. — https://pubmed.ncbi.nlm.nih.gov/31103085/
- See also: Ultrasonographic quantification of intrinsic hand muscle cross-sectional area; reliability and validity for predicting muscle strength — https://pubmed.ncbi.nlm.nih.gov/25482051/